CLINICAL TRIAL: NCT01826370
Title: A Post-Marketing Surveillance Study on the Safety, Tolerability and Efficacy of Linagliptin Among Filipino Patients With Type 2 Diabetes Mellitus
Brief Title: Linagliptin Among Filipino Patients With Type 2 Diabetes Mellitus
Status: Terminated | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1218.94
Record Dates: First submitted 2013-04-04; First posted 2013-04-08 (Estimated); Results first posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Linagliptin
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: Linagliptin — tablet

SUMMARY:
This is a prospective, non-interventional, open label, multi center, post marketing surveillance study designed to assess the safety, tolerability and efficacy of Linagliptin among Filipino patients with type 2 Diabetes Mellitus (DM) within the study duration of 24 weeks.

ELIGIBILITY:
Inclusion criteria:

1. Filipino of Asian race
2. Patient using Linagliptin within label or locally approved indication. The prescription of Linagliptin to the patient must be in the course of normal clinical practice and independent of the decision to include the patient in the study.
3. Male or female patients more than 18 years old
4. Body mass index less than or equal to 40
5. Diagnosed with type 2 DM
6. Uncontrolled type 2 DM with fasting blood sugar of more than 126 mg/dl and/or HbA1c more than 7%.

Exclusion criteria:

1. Diagnosed with type 1 DM
2. Patients with acute illness requiring hospitalization in the past one month
3. Patients participating in a different study that includes an investigational drug
4. Patients with known hypersensitivity reaction to Linagliptin or any of tis components
5. Pregnant women and those women who have intentions of getting pregnant within the study duration
6. Nursing women
7. Patients with concomitant conditions that contraindicates Linagliptin use as described in its product information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Filipino type 2 DM patients
Sampling Method: Non-Probability Sample
Enrollment: 678 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (51):
- Philippines (51):
  - Boehringer Ingelheim Investigational Site 43, Agoo, La Union
  - Boehringer Ingelheim Investigational Site 40, Angeles City, Pampanga
  - Boehringer Ingelheim Investigational Site 31, Angono, Rizal
  - Boehringer Ingelheim Investigational Site 32, Antipolo, Rizal
  - Boehringer Ingelheim Investigational Site 27, Aparri, Cagayan
  - Boehringer Ingelheim Investigational Site 4, Batangas
  - Boehringer Ingelheim Investigational Site 48, Butuan City, Agusan Del Norte
  - Boehringer Ingelheim Investigational Site 12, Cabanatuan, Nueva Ecija
  - Boehringer Ingelheim Investigational Site 23, Cagayan de Oro
  - Boehringer Ingelheim Investigational Site 3, Caloocan
  - Boehringer Ingelheim Investigational Site 42, Cardona, Rizal
  - Boehringer Ingelheim Investigational Site 25, Cebu
  - Boehringer Ingelheim Investigational Site 44, Dagupan, Pangasinan
  - Boehringer Ingelheim Investigational Site 49, Iligan City, Lanao Del Norte
  - Boehringer Ingelheim Investigational Site 2, Iloilo City
  - Boehringer Ingelheim Investigational Site 45, Iriga City, Camarines Sur
  - Boehringer Ingelheim Investigational Site 20, Laoag, Ilocos Norte
  - Boehringer Ingelheim Investigational Site 24, Las Piñas
  - Boehringer Ingelheim Investigational Site 7, Legazpi, Albay
  - Boehringer Ingelheim Investigational Site 35, Lucena, Quezon
  - Boehringer Ingelheim Investigational Site 1, Makati
  - Boehringer Ingelheim Investigational Site 39, Malolos, Bulacan
  - Boehringer Ingelheim Investigational Site 37, Mandaluyong
  - Boehringer Ingelheim Investigational Site 28, Manila
  - Boehringer Ingelheim Investigational Site 5, Marikina City
  - Boehringer Ingelheim Investigational Site 16, Meycauyan, Bulacan
  - Boehringer Ingelheim Investigational Site 47, Naga City, Camarines Sur
  - Boehringer Ingelheim Investigational Site 15, Olongapo City
  - Boehringer Ingelheim Investigational Site 10, Pampanga
  - Boehringer Ingelheim Investigational Site 19, Paranaque City
  - Boehringer Ingelheim Investigational Site 51, Pasay
  - Boehringer Ingelheim Investigational Site 30, Pasig
  - Boehringer Ingelheim Investigational Site 34, Puerto Princesa, Palawan
  - Boehringer Ingelheim Investigational Site 26, Quezon City
  - Boehringer Ingelheim Investigational Site 11, Rosales, Pangasinan
  - Boehringer Ingelheim Investigational Site 21, San Fernando, La Union
  - Boehringer Ingelheim Investigational Site 9, San Fernando, Pampanga
  - Boehringer Ingelheim Investigational Site 13, San Jose, Nueva Ecija
  - Boehringer Ingelheim Investigational Site 29, San Juan City
  - Boehringer Ingelheim Investigational Site 8, San Pablo, Laguna
  - Boehringer Ingelheim Investigational Site 50, San Pedro, Laguna
  - Boehringer Ingelheim Investigational Site 41, Santiago City, Isabela
  - Boehringer Ingelheim Investigational Site 36, Sogod, Southern Leyte
  - Boehringer Ingelheim Investigational Site 38, Sta.Maria, Bulacan
  - Boehringer Ingelheim Investigational Site 6, Tacloban City
  - Boehringer Ingelheim Investigational Site 33, Tagbilaran, Bohol
  - Boehringer Ingelheim Investigational Site 14, Tuguegarao, Cagayan
  - Boehringer Ingelheim Investigational Site 18, Urdaneta, Pangasinan
  - Boehringer Ingelheim Investigational Site 46, Valencia City Bukidnon
  - Boehringer Ingelheim Investigational Site 17, Valenzuela, Bulacan
  - Boehringer Ingelheim Investigational Site 22, Zamboanga City

RESULTS

PARTICIPANT FLOW:
Groups:
- Linagliptin: Linagliptin 5 mg was administered orally once a day for 24 weeks
Period: Overall Study
Arm/Group | Linagliptin
Started | 678
Completed | 658
Not Completed | 20
Not completed — Protocol Violation | 6
Not completed — Lost to Follow-up | 12
Not completed — Other reason not defined above | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set which consisted of all patients who have taken at least one dose of linagliptin and participated in the follow-up visit, thus, having a baseline and end-point evaluation.
Arm/Group | Linagliptin
Number analyzed (Participants) | 660
Age, Continuous [Mean (Standard Deviation); unit: years] — Age information is missing for 5 patients
  years | 57.67 (13.3)
Gender [Number; unit: participants] — Gender information is missing for 4 patients
  participants
    Female | 360
    Male | 296

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events and Serious Adverse Events
Description: Frequency of adverse events and serious adverse events in an actual clinical setting, including hypoglycemic events.
Time Frame: Week 24
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Linagliptin
Number analyzed (Participants) | 660
percentage of participants
  Adverse Events | 0.8
  Serious Adverse Events | 0.0

2. Secondary Outcome: Change From Baseline to Week 24 of HbA1c
Description: Change from baseline to week 24 of glycosylated hemoglobin (HbA1c)
Time Frame: Baseline and 24 weeks
Population: Effectiveness analysis set which included patients with complete baseline and follow up secondary outcomes. For this outcome measure this include patients with baseline and end-point data for HbA1c.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Linagliptin
Number analyzed (Participants) | 625
percentage of HbA1c | -1.7 (1.5)

3. Secondary Outcome: Change From Baseline to Week 24 of Fasting Blood Sugar
Description: Change from baseline to week 24 of fasting blood sugar
Time Frame: Baseline and 24 weeks
Population: Effectiveness analysis set which included patients with complete baseline and follow up secondary outcomes. For this outcome measure this include patients with baseline and end-point data for fasting blood sugar.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Linagliptin
Number analyzed (Participants) | 629
mg/dl | -65.0 (66.5)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Safety analysis set which consisted of all patients who have taken at least one dose of linagliptin and participated in the follow-up visit, thus, having a baseline and end-point evaluation.
Arm/Group | Linagliptin
Serious Adverse Events (participants affected / at risk) | 0/660
Other Adverse Events (participants affected / at risk) | 0/660

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.